CLINICAL TRIAL: NCT03334175
Title: Walnuts to Achieve Lasting NUTrition to Prevent Diabetes (WALNUT-Diabetes)
Brief Title: Walnuts to Achieve Lasting NUTrition to Prevent Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4000-128070-125731P-44
Record Dates: First submitted 2017-10-30; First posted 2017-11-07 (Actual); Results first posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: PreDiabetes; Overweight and Obesity
MeSH Terms: conditions — Prediabetic State; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Walnuts Now (Experimental): Will receive and be instructed to consume 1-oz individually wrapped daily walnut supplement packages for 12 weeks during intervention.
  Interventions: Drug: Walnuts
- Walnuts Later (No Intervention): Will receive diet and exercise guidance at beginning of study. At end of study, will receive 12 weeks of a walnut supply to be consumed at their discretion after the study is complete.

INTERVENTIONS:
Drug: Walnuts — 1 ounce of individually wrapped, raw walnuts to be consumed daily replacing a high-refined carbohydrate food.
  Arms: Walnuts Now

SUMMARY:
Prediabetes is a precursor of type 2 diabetes and an independent risk factor for cardiovascular disease, and currently affects one-quarter of the population of the United States. Individuals of overweight or obese BMI are at particular high risk for incident diabetes. A major modifiable risk factor for type 2 diabetes is poor dietary quality, and improvement of dietary quality can effectively delay and even prevent type 2 diabetes. Interventions to improve dietary quality thus far, however, rely on short-term intensive clinically designed meals replacing the entire diet which have poor sustainability. Persistent improvements to daily dietary patterns are often difficult without directed guidance, and overall dietary quality in the United States remains poor. The identification of a practical, daily dietary intervention to improve dietary quality and prevent diabetes in those at high risk remains unknown. The investigators propose to enroll 40 individuals with diagnosed prediabetes into a randomized controlled pilot study and provide a daily walnut supplementation intervention to determine feasibility and acceptability of the supplement. The investigators will then determine preliminary efficacy on metabolic markers and will investigate associations between dietary quality and circulating levels of branched-chain amino acids. The goal is to implement a whole-food supplement to improve dietary quality in patients with prediabetes as a tool for future type 2 diabetes prevention.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18-65 years of age at baseline living in the San Francisco Bay area.
2. BMI>25 m/kg2 (or >23 m/kg2 for individuals of Asian or South Asian ethnicity)
3. Documentation of prediabetes diagnosis as evidenced by the following criteria:

   1. A fasting glucose 100-125 mg/dL, or a HbA1c measurement of 5.7-6.4%, OR a diagnosis of "prediabetes" or "impaired fasting glucose" in the past 6 months, identified through an electronic medical record query from patients at UCSF and through outside recruitment in the surrounding community
   2. We will confirm eligibility of potential participants by repeating fasting capillary blood glucose measurements at the baseline visit to ensure that they have prediabetes
4. Written informed consent and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Pregnant or breastfeeding women at enrollment.
2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data, such as diverticulosis or diverticulitis.
3. Tree or peanut allergies
4. Unwilling to consume a daily walnut supplement.
5. Diagnosis of diabetes
6. On glucose lowering medications
7. Dietician-managed dietary intake, or personal or medical dietary restrictions that do not allow consumption of walnuts
8. Malabsorptive conditions including intestinal bypass surgery, pancreatitis, inflammatory bowel disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meghana Gadgil, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Walnuts Now | Walnuts Later
Started | 8 | 10
Completed | 8 | 9
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Walnuts Now | Walnuts Later | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Continuous [Mean (Full Range); unit: years] | 55.4 [47 to 62] | 57.1 [32 to 65] | 56.3 [32 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 6 | 5 | 11
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 10 | 18
Fasting glucose [Mean (Standard Deviation); unit: mg/dL] | 109.5 (24.6) | 106 (11.5) | 107.6 (17.9)
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage of Hemoglobin A1c] | 5.8 (0.8) | 5.9 (0.3) | 5.9 (0.6)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.4 (4.1) | 35.6 (5.9) | 33 (5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Recruited and Retained
Description: Number of participants recruited and retained
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Walnuts Now | Walnuts Later
Number analyzed (Participants) | 8 | 10
Participants | 8 | 9

2. Primary Outcome: Adherence to the Intervention
Description: Adherence to the intervention was determined through daily food diaries. Participants detailed daily consumption of the walnut supplement on a calendar provided at the outset of the study. Percentage was determined as number of days consuming supplement over 84 days total.
Time Frame: 12 weeks
Population: Adherence was not measured in the control group who did not receive the walnut supplement.
Measure: Mean (Full Range); unit: percentage of days
Arm/Group | Walnuts Now | Walnuts Later
Number analyzed (Participants) | 8 | 0
percentage of days | 74.7 [47 to 93] |

3. Primary Outcome: Palatability of Supplement
Description: Palatability was measured using a visual analog scale, the scale range is 0-100, with 100 being the "Most Pleasant."
Time Frame: 12 weeks
Population: Palatability was not measured in the control group who did not receive the walnut supplement intervention.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Walnuts Now | Walnuts Later
Number analyzed (Participants) | 8 | 0
score on a scale | 87 [70 to 100] |

4. Secondary Outcome: Change in Diet Quality
Description: Change in diet quality measured by Healthy Eating Index-2010 Score (0 - 100). Higher scores indicate better diet quality.
Time Frame: 0 weeks and 12 weeks
Population: The "Walnuts Later" group did not complete the food frequency questionnaire required to assess change in diet quality. As the primary outcome was feasibility of recruitment and retention, we chose to analyze diet quality data only in those participants who provided these data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Walnuts Now | Walnuts Later
Number analyzed (Participants) | 8 | 6
score on a scale | 2.1 (11.9) | 2.9 (6.2)

5. Secondary Outcome: Fasting Glucose
Description: Change in fasting glucose
Time Frame: 0 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Walnuts Now | Walnuts Later
Number analyzed (Participants) | 8 | 9
mg/dL | -4.75 (9.8) | 1.2 (7.5)

6. Secondary Outcome: Change in Hemoglobin A1c
Description: Change in percentage of Hemoglobin A1c
Time Frame: 0 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of A1c
Arm/Group | Walnuts Now | Walnuts Later
Number analyzed (Participants) | 8 | 9
percentage of A1c | -0.05 (0.13) | -0.08 (0.21)

7. Secondary Outcome: Change in Low Density Lipoprotein Levels
Description: Change in low density lipoprotein levels from baseline to 12 weeks
Time Frame: 0 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Walnuts Now | Walnuts Later
Number analyzed (Participants) | 8 | 9
mg/dL | -8.4 (15.5) | -0.5 (13.1)

8. Other Pre Specified Outcome: Number of Participants Who Had Plasma Metabolomics Performed
Description: Plasma metabolomics performed as an exploratory outcome for all participants. This outcome represents number of participants who had a successful blood draw at both baseline and 12 weeks sent to the laboratory with usable data recovered.
Time Frame: 0 weeks and 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Walnuts Now | Walnuts Later
Number analyzed (Participants) | 8 | 9
Participants | 8 | 9

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Walnuts Now | Walnuts Later
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT03334175/Prot_SAP_001.pdf